CLINICAL TRIAL: NCT01485510
Title: Evaluation of the New Orleans Intervention for Infant Mental Health in Glasgow
Brief Title: Evaluation of the New Orleans Intervention for Infant Mental Health
Acronym: BEST?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Helen Minnis, Principal Investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CZH/4/629
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Maltreated Infants
Keywords: Maltreatment; Infant Mental Health; Infant mental health in maltreated children
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glasgow Infant and Family Team (GIFT) (Experimental): A service developed by Charles Zeanah and colleagues in New Orleans, that aims to improve the mental health of maltreated infants.
  Interventions: Behavioral: GIFT
- Family Assessment & Contact Service (Active Comparator): A social-work based service that aims to assess maltreated children and make recommendations about their future care.
  Interventions: Behavioral: FACS

INTERVENTIONS:
Behavioral: GIFT — An attachment-based assessment, then a tailored intervention aimed at maximising the chances of a maltreated child returning to the birth family.
  Other Names: New Orleans Intervention
  Arms: Glasgow Infant and Family Team (GIFT)
Behavioral: FACS — A social work assessment of family functioning that makes recommendations regarding future placement of a maltreated child.
  Other Names: Case Management (Lieberman, 2005).
  Arms: Family Assessment & Contact Service

SUMMARY:
Early intervention for maltreated infants can improve mental and physical health throughout life and benefit families and society as a whole. The New Orleans Model provides intensive assessment and treatment for families of maltreated preschool children in foster care, with recommendations to court about adoption, or permanent return to birth families. The New Orleans Model appears to have led to better informed decisions about permanent placement and to better child mental health in Louisiana. The investigators propose an exploratory randomised controlled trial investigating the effectiveness of the New Orleans Model in the Scottish context, informing the development of an economic model to explore the potential cost-effectiveness. Families with a maltreated child under 5 years of age will be offered the New Orleans Model or "case management" i.e. quality assured services as usual, using random allocation. The investigators will measure outcome using well validated measures of parent-child interaction, cognition and attachment.

DETAILED DESCRIPTION:
The first 5 months of this trial - from December 2011 to April 2012 - is an internal pilot or "implementation period". During this time we have fewer research staff, both services will just have started and we will only be collecting selected outcome measures. These will be the Principle Outcome Measure, the Infant-Toddler Social-Emotional Assessment (ITSEA), plus the Disturbance of Attachment Interview (DAI) and Parent-Infant Global Assessment of Functioning (PIR-GAS). We hope to include data from implementation period in our trial analysis, but if results are very different due to services "bedding in", we may not do so

ELIGIBILITY:
Inclusion Criteria:

* All maltreated children placed in foster care, aged between 6 and 60 months, whose parents give informed opt-in consent

Exclusion Criteria:

* Children with profound learning disability

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 227 (Actual)
Dates: Start 2011-12; Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Change in score on the Infant-Toddler Social-emotional Assessment (ITSEA) | Baseline and at 1 year follow-up
  The ITSEA is a well validated parent/carer-completed questionnaire covering a wide range of social and emotional behaviours in infants and preschool children. It has been shown to be sensitive to change in previous intervention research with maltreated children with medium to large effect sizes and has good longitudinal stability.

SECONDARY OUTCOMES:
The Parent Evaluation of Development (PEDS) | Baseline and 1 year follow up
  A brief parent-report measure of infant language and other milestones
The Disturbances of Attachment Interview (DAI) | Baseline and 1 year follow up
  A measure of attachment disorder.
The Parent-Infant Global Assessment of Functioning (PIR-GAS) | Baseline and 1 year follow up
  A video-based assessment of global relationship functioning
This is My Baby (TIMB) | Baseline and 1 year Follow up
  A measure of the degree of committment to the child by the caregiver
The Development and Wellbeing Assessment (DAWBA) | Baseline and 1 year follow up for children over 2 years.
  A diagnostic intrument generating DSM and ICD psychiatric diagnoses.
Cognitive assessment | Baseline and 1 year follow up
  This will be either the Bayley's or the WPPSI depending on the age of the child.
The Use of Services Questionnaire | Baseline and 1 year follow up
  This carer-report questionnaire generates service use and costs data for health economic analysis
The Strange Situation Procedure (SSP) | 1 year follow up only
  This is the gold standard measure for infant/toddler attachment patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Minnis, MBChB, PhD, Principal Investigator — University of Glasgow; Niel Campbell, MBChB, PhD, Study Chair — University of Aberdeen
Locations (1):
- University of Glasgow, Glasgow, United Kingdom